CLINICAL TRIAL: NCT04307355
Title: Evaluation of Oxygen Delivery With TransCu O2 to Study Success Rate of Surgically Closed Wounds
Brief Title: Continuous Diffusion of Oxygen Treatment for Incision Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Electrochemical Oxygen Concepts, Inc. (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-46332
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Surgical Wound; Breast Surgery; Mammoplasty; Incision Wound
Keywords: Infection; Dehiscense; Tissue infection; Surgical Revision; Scar tissue; Wound Closure
MeSH Terms: conditions — Surgical Wound; Infections; Cicatrix

STUDY DESIGN:
Intervention Model Description: Each participant will act as their own control in this model. One of the participant's breasts will receive the intervention dressing while the other intervention breast will receive the standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Direct Continuous Diffusion of Oxygen (dCDO) (Active Comparator): One of the participant's breasts will be provided with a Transcu O2 ® Oxygen delivery system and 4x4 dressing at the surgical site for 4 weeks as supportive care. The 4x4 dressing will be attached to breast using Tegaderm adhesive.
  Interventions: Device: Transcu O2®; Other: Tegaderm
- Control (No Intervention): One of the participant's breasts will receive a standard-of-care at the surgical site and will be followed for 4 weeks.
- Silicon Continuous Diffusion of Oxygen (sCDO) (Active Comparator): One of the participant's breasts will be provided with a Transcu O2 ® Oxygen delivery system and 4x4 dressing at the surgical site for 4 weeks as supportive care. The 4x4 dressing will be attached to breast using Silagen adhesive.
  Interventions: Device: Transcu O2®; Other: Silagen

INTERVENTIONS:
Device: Transcu O2® — Breasts randomized into study active group will be provided with a Transcu O2® at their surgical site and followed for 4 weeks.
  Arms: Direct Continuous Diffusion of Oxygen (dCDO); Silicon Continuous Diffusion of Oxygen (sCDO)
Other: Tegaderm — A 10 cm × 12 cm Tegaderm TM Film adhesive (3M Healthcare, Minnesota).
  Arms: Direct Continuous Diffusion of Oxygen (dCDO)
Other: Silagen — A 10 cm × 12 cm silicon sheet (Silagen, New Medical Technology, Inc, Illinois).
  Arms: Silicon Continuous Diffusion of Oxygen (sCDO)

SUMMARY:
This is an exploratory randomized controlled trial study to test feasibility, acceptability, and proof of concept efficacy of Continuous Diffusion of Oxygen (CDO) adjunct therapy for decreasing healing time and reducing tissue necrosis post breast reconstruction. The investigator will assess the benefit of this novel adjunct therapy on successful closure, tissue oxygenation, scar appearance, and patients centered outcomes including perception of benefit, pain, sleep quality, and quality of life.

Eligible subjects will be randomly (ratio 1:1) assigned to either intervention group (IG) or control group (CG) and will be followed for four weeks. Both groups will receive standard of care for wound treatment. IG will also receive CDO adjunct therapy using a novel dressing, which facilitates continuously supplies oxygen to the wound inside the wound dressing using a portable device named TransCu O2.

The study device TransCu O2® is a Class II medical device which has US Food and Drug Administration (FDA) 510(k) clearance, CE-Mark approval and a Health Canada license for the treatment of wounds. Outcomes will be assessed on weekly-basis up to 4 weeks.

DETAILED DESCRIPTION:
Surgical wound complications such as infection, dehiscence, necrotic tissue, surgical revision, and poor cosmesis are unfortunately highly prevalent in patients post breast reconstruction. In particular, necrosis/ischemia post breast reconstruction because of poor blood circulation is highly prevalent and is estimated to be occurring in up to 75% of cases leading to excessive scar formation. Some factors such as active smoking or an underlying disease such as diabetes and history of radiation therapy could increase the likelihood of excessive scar and/or necrosis.

In most cases surgical wounds are managed with a simple island dressing, wool padding and a light retention bandage. It could be argued that such low cost, traditional dressings are adequate for most surgical wounds. However, patients with poor tissue blood circulation often require modern wound care products that offer additional benefits, in particular among those with vascular and poor tissue oxygenation problem. Poor tissue oxygenation and poor skin perfusion could lead to surgical wound complications such as wound inflection, tissue necrosis, pain, trauma and untimely surgical revision. In particular, the presence of non-viable necrotic tissue is significant as it can be responsible for delaying healing, prolonging the inflammatory response, mechanically obstructing contraction and impeding re-epithelialisation. It also provides a focus for wound infection and surgical revision.

Even after successful healing, necrotic tissue could still lead to excessive scar formation. Many of these scars can be problematic, being aesthetically unpleasant and causing discomfort. Blood supply is a significant factor in wound healing, and area of the skin with rich supply of vasculature is known to heal with finer scars. Several studies have demonstrated that mild hypoxia (lack of transcutaneous oxygen) is present in early scars, moderate hypoxia in proliferative scars, and severe hypoxia in regressive scars. Oxygen levels then return to normal in mature scars, which is consistent along with the dynamic change in microvessel density. Therefore level of transcutaneous oxygen could be a determinant factor in formation of excessive scar formation.

Continuous Diffusion of Oxygen (CDO) is a treatment modality that delivers pure oxygen to wounds using the same basic mechanism as breathing, namely direct diffusion into the wound from a moist surface. Because impaired blood flow results in impaired oxygen supply to incisional wounds, investigators have researched the potential of oxygen saturation, or supersaturation, to reinitiate or even accelerate wound healing. Oxygen has been shown to result in not only faster wound closure, yet also better strength of repair and higher organization of collagen, which in turn can result in lower wound recidivism and better scar appearance.

In this feasibility and proof of concept study, The investigator plan to investigate the effects of oxygen on incisional wound repair and scarring after mastectomy and breast reconstruction. The investigator will use a device (TransCu O2® Oxygen Delivery System ) which continuously supplies oxygen to the wound inside the wound dressing. The device the investigator used, the TransCu O2 System, (EO2 Concepts®, San Antonio, TX) is small, wearable and silent. The system is FDA-approved and CDO therapy has been the subject of a growing body of clinical experience and scientific investigations demonstrating good results. The therapy is similar in theory to the intermittent application of oxygen through Hyperbaric Oxygen (HBO) and Topical Oxygen (TO), with a few key differences summarizing in the following:

1) CDO provides continuous therapy, providing ~twenty-fold longer time of oxygen delivery versus intermittent therapies that are only applied 90 minutes a day. 2) CDO allows for full patient mobility during treatment, thereby reducing the risk of non-compliance and reducing overall costs

The investigator have successfully used CDO therapy to reduce likelihood of tissue necrosis after surgical closure post lower extremity amputation as well as post parathyroid surgery, in which over 20 subjects were recruited and no adverse outcomes were reported. The investigator plan to extend our study to determine whether CDO therapy would show decreased healing time and better scar cosmesis early on for standardized incisional wounds such as breast reconstruction. The investigator hypothesis that using CDO will reduce the likelihood of necrotic tissue as well as severe incisional scar post-surgical closure by improving transcutaneous oxygen levels during wound healing process. The investigator will examine the validity of this hypothesis using a pilot randomized controlled trial using a convenient sample of 40 people (20 subjects per arm) after mastectomy and breast reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years of age
* Ability to provide informed consent
* Presence of a wound due to surgical intervention and closure
* Subject or responsible caregiver is willing and able to maintain the required Continuous Diffusion of Oxygen (CDO) system (if assigned to the intervention group) and applicable dressing changes

Exclusion Criteria:

* Active Drug/alcohol abuse (or history of drug/alcohol abuse in last 1 month)
* Dementia or severely impaired cognitive function
* excessive lymphedema
* presence of active infection
* subject has a history of or any intercurrent illnesses or conditions that would compromise the safety of the subject according to judgement of a qualified wound specialist

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Najafi, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Baylor College of Medicine's Plastic Surgery Department through surgeon referrals or chart reviews. Of the 23 participants who met the inclusion criteria and enrolled, 3 withdrew.
Pre-assignment Details: Surgeries were performed on both breasts, with the intervention randomized to either the left or right breast, while the contralateral side served as the control. In other words, each subject acted as their own control. This resulted in data from 40 breasts across 20 participants-20 control and 20 intervention.
Units Other Than Participants: Breasts
Groups:
- Direct CDO (dCDO): Participants will be provided with a Transcu O2 ® Oxygen delivery system at the surgical site for 4 weeks as supportive care.
  One of the participant's breasts will be provided with a Transcu O2 ® Oxygen delivery system and 4x4 dressing at the surgical site for 4 weeks as supportive care. The 4x4 dressing will be attached to breast using Tegaderm adhesive.
- Control: Participants will be placed in a standard dressing at the surgical site and will be followed for 4 weeks.
- Silicon CDO (sCDO): One of the participant's breasts will be provided with a Transcu O2 ® Oxygen delivery system and 4x4 dressing at the surgical site for 4 weeks as supportive care. The 4x4 dressing will be attached to breast using Silicon sheet.
Period: Overall Study
Arm/Group | Direct CDO (dCDO) | Control | Silicon CDO (sCDO)
Started (Please note that the total number of participants was 23, of whom 3 withdrew. Surgeries were performed on both breasts, with the intervention (either dCDO or sCDO) randomized to the left or right breast, while the contralateral side served as the control. In other words, each subject acted as their own control. This design resulted in data from 40 breasts across 20 participants: 20 control breasts and 20 intervention breasts (10 dCDO and 10 sCDO).) | 13; 13 Breasts | 23; 23 Breasts | 10; 10 Breasts
Completed (Surgeries were performed on both breasts, with the intervention (either dCDO or sCDO) randomized to either the left or right breast, while the contralateral side served as the control. This design included 10 participants receiving dCDO and 10 receiving sCDO, with the contralateral breast of all 20 participants serving as the control. Unfortunately, ClinicalTrials.gov automatically calculates the total number of participants as double the actual count in this case) | 10; 10 Breasts (Surgeries were performed on both breasts, with the intervention randomized to either the left or right breast, while the contralateral side served as the control for each intervention arm. Therefore, in this context, the "units" refer to individual "breasts.") | 20; 20 Breasts | 10; 10 Breasts
Not Completed | 3; 3 Breasts | 3; 3 Breasts | 0; 0 Breasts
Not completed — Non-Compliance | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants are counted as individual breasts, with one breast treated with the intervention and the other with the standard of care. The study included 20 participants, resulting in 20 control breasts from 20 participants. Of the intervention breasts, 10 participants received dCDO and 10 received sCDO.
Units Other Than Participants: Breasts
Groups:
- Direct CDO (dCDO): One of the participant's breasts will be provided with a Transcu O2 ® Oxygen delivery system and 4x4 dressing at the surgical site for 4 weeks as supportive care. The 4x4 dressing will be attached to breast using Tegaderm adhesive.
- Silicone CDO (sCDO): One of the participant's breasts will be provided with a Transcu O2 ® Oxygen delivery system and 4x4 dressing at the surgical site for 4 weeks as supportive care. The 4x4 dressing will be attached to breast using silicon sheet.
- Total: Total of all reporting groups
Arm/Group | Direct CDO (dCDO) | Control | Silicone CDO (sCDO) | Total
Number analyzed (Participants) | 10 | 20 | 10 | 20
Number analyzed (Breasts) | 10 | 20 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Surgeries were performed on both breasts, with the intervention randomized to either the left or right breast, while the contralateral side served as the control for each intervention arm. Since each subject acted as their own control, there were no differences in age or other demographic factors between the control arms and the total cases.
  years | 32.70 (6.02) | 34.45 (10.56) | 38.20 (13.34) | 34.45 (10.33)
Sex/Gender, Customized [Number; unit: participants]
  Female | 10 | 20 | 10 | 20
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Each breast was treated as an independent sample. For each participant, one breast was randomly designated as the control, while the other was assigned to one of the two intervention groups: sCDO or dCDO. Consequently, the number of cases in the ethnicity category was duplicated
  participants
    Black or African American | 9 | 18 | 9 | 18
    White | 1 | 2 | 1 | 2
Region of Enrollment [Number; unit: participants] — Population: Only the participants who completed the study where included for analysis.
  participants
    United States | 10 | 20 | 10 | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Only the participants who completed the study where included for analysis.
  kg/m^2 | 32.92 (6.18) | 34.27 (5.29) | 35.61 (4.30) | 34.27 (5.29)

OUTCOME MEASURES:

1. Primary Outcome: Wound Size at 4 Weeks
Description: Wound size will be traced and quantified using a wound imaging system (Snapshot, Kent Imaging)
Time Frame: 4 weeks
Population: Baseline participants are counted as individual breasts, with one breast treated with the intervention and the other with the standard of care. The study included 20 participants, resulting in 20 control breasts. Of the intervention breasts, 10 received dCDO and 10 received sCDO.
Measure: Mean (Standard Deviation); unit: cm^2
Units Other Than Participants: Breasts
Arm/Group | Direct Continuous Diffusion of Oxygen (dCDO) | Control | Silicon Continuous Diffusion of Oxygen (sCDO)
Number analyzed (Participants) | 10 | 20 | 10
Number analyzed (Breasts) | 10 | 20 | 10
cm^2 | 1.5 (2.83) | 2.75 (7.2) | 0.15 (0.06)

2. Primary Outcome: Incidence of Wound Complication at 4 Weeks
Description: Complication is described as infection, dehiscence, and/or necrotic tissue
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Units; unit: Breasts
Units Other Than Participants: Breasts
Arm/Group | Direct Continuous Diffusion of Oxygen (dCDO) | Control | Silicon Continuous Diffusion of Oxygen (sCDO)
Number analyzed (Participants) | 10 | 20 | 10
Number analyzed (Breasts) | 10 | 20 | 10
Breasts | 1 | 3 | 0

3. Secondary Outcome: Presence of Scar Tissue
Description: Scar tissue presence will be assessed by simple view.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Units; unit: Breasts
Units Other Than Participants: Breasts
Arm/Group | Direct Continuous Diffusion of Oxygen (dCDO) | Control | Silicon Continuous Diffusion of Oxygen (sCDO)
Number analyzed (Participants) | 10 | 20 | 10
Number analyzed (Breasts) | 10 | 20 | 10
Breasts | 0 | 0 | 0

4. Secondary Outcome: Change in DeoxyHB From Baseline to 4 Weeks
Description: DeoxyHb at the T-Junction of each breast will be assessed using near-infrared spectroscopy (Snapshot, Kent Imaging). DeoxyHb is measured as a fraction ranging from 0 to 1. The reported values below are the estimate percent change from the baseline visit to the 4th week visit.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Error); unit: percentage change
Units Other Than Participants: Breasts
Arm/Group | Direct Continuous Diffusion of Oxygen (dCDO) | Control | Silicon Continuous Diffusion of Oxygen (sCDO)
Number analyzed (Participants) | 10 | 20 | 10
Number analyzed (Breasts) | 10 | 20 | 10
percentage change | 83.89 (15.89) | 136.07 (23.28) | 46.53 (25.698)

5. Secondary Outcome: Self-reported Pain at Week 4
Description: Pain will be assessed with visual analogue scale from 0 to 10 where 10 is the worst pain ever. At the final visit, patients were asked to rate their pain on this scale using the POSAS (Patient and Observer Scar Assessment Scale) questionnaire. An average of this score was taken across each group.
Time Frame: At 4 weeks
Population: The pain questionnaire was not asked until the sCDO group was added. Therefore, 0 samples from the dCDO group were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Direct Continuous Diffusion of Oxygen (dCDO) | Control | Silicon Continuous Diffusion of Oxygen (sCDO)
Number analyzed (Participants) | 0 | 6 | 9
units on a scale |  | 2.3 (2.8) | 3.9 (2.75)

6. Secondary Outcome: Change in Tissue Oxygen Saturation (SatO2) From Baseline to 4 Weeks
Description: SatO2 at the T-Junction of each breast will be assessed using near-infrared spectroscopy (Snapshot, Kent Imaging). SatO2 is measured as a fraction ranging from 0 to 1. The reported values below are the estimate percent change from the baseline visit to the 4th week visit.
Time Frame: Baseline to 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage change
Units Other Than Participants: Breasts
Arm/Group | Direct Continuous Diffusion of Oxygen (dCDO) | Control | Silicon Continuous Diffusion of Oxygen (sCDO)
Number analyzed (Participants) | 10 | 20 | 10
Number analyzed (Breasts) | 10 | 20 | 10
percentage change | -33.57 (5.84) | -23.30 (5.82) | 13.76 (12.12)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study duration, up to 4 weeks for each participant.
Arm/Group | Direct Continuous Diffusion of Oxygen (dCDO) | Control | Silicon Continuous Diffusion of Oxygen (sCDO)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 2/20 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct Continuous Diffusion of Oxygen (dCDO) (N=10) | Control (N=20) | Silicon Continuous Diffusion of Oxygen (sCDO) (N=10)
Allergy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Skin allergy to Tegarderm adhesive
Skin irritation (Non-study related) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Non-study related skin irritation in both breasts
Itching, mild breakdown, and drainage (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Participant removed the dressing for 10 days and then re-applied

LIMITATIONS AND CAVEATS:
Surgeries were performed on both breasts, with the intervention (either dCDO or sCDO) randomized to either the left or right breast, while the contralateral side served as the control. This design included 10 participants receiving dCDO and 10 receiving sCDO, with the contralateral breast of all 20 participants serving as the control. Unfortunately, ClinicalTrials.gov automatically calculates the total number of participants as double the actual count in this case.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04307355/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04307355/ICF_001.pdf